CLINICAL TRIAL: NCT04860518
Title: A Phase II Multi-Center, Double-Blind, Randomized and Controlled Study of the Safety and Efficacy of Intravenous Recombinant Human Interferon Beta-1a in Comparison to Dexamethasone for the Treatment of Hospitalized Patients With COVID-19 Infection
Brief Title: Human Intravenous Interferon Beta-Ia Safety and Preliminary Efficacy in Hospitalized Subjects With COVID-19
Acronym: HIBISCUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision is based on changes in the pandemic and further weakening of the recruitment that will not enable a completion of the study in any reasonable time
Sponsor: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FP1CLI017
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Results first posted 2022-10-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — peginterferon beta-1a; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be performed in a double-blind and randomized manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV IFN beta-1a (Experimental): Patients receiving active drug: will receive two separate bolus injections one containing IFN-beta -1a and another injection containing Saline.
  Interventions: Drug: IFN beta-1a
- IV Dexamethasone (Active Comparator): Patients receiving active comparator: will receive two separate bolus injections one containing saline and another injection containing Dexamethasone.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: IFN beta-1a — Treated daily with IFN beta-1a 10 μg as an IV bolus for 6 days while hospitalised
  Arms: IV IFN beta-1a
Drug: Dexamethasone — Treated daily with dexamethasone 6 mg as an IV bolus for 6 days while hospitalised
  Arms: IV Dexamethasone

SUMMARY:
This double-blinded, randomized study is being conducted to see if the investigational new drug called FP-1201-lyo - intravenous Interferon beta-1a, hereafter IV IFN beta-1a, can help patients recover more quickly from COVID-19 and prevent worsening of the condition. To understand if IV IFN beta-1a can help treat patients with COVID-19, this study drug will be compared to dexamethasone.

Study subjects will be treated daily with IV IFN beta-1a 10 μg or IV dexamethasone for 6 consecutive days while hospitalized and will undergo daily assessments while in hospital for a maximum of 28 days. Study specific assessments will be collected at pre-dose Day 1 through Day 28 (PD and PIM assessments), in addition, clinical routine assessments will be utilized for safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Positive SARS-CoV-2 test by PCR (polymerase chain reaction) or other diagnostic method within the past 7 days
3. Admission to hospital with respiratory symptoms of COVID-19 requiring hospital care and oxygen supplementation (≤ 8L/min)
4. Respiratory symptom onset no more than 7 days prior to hospital arrival
5. Informed consent from the subject or the subject's personal legal representative or a professional legal representative must be available

Exclusion Criteria:

1. Unable to screen, randomize and administer study drug within 48 hours from arrival to hospital
2. Systemic corticosteroid, baricitinib or tofacitinib (or other JAK-STAT signalling pathway inhibitors) therapy within 7 days prior to arrival to hospital or planned for the next days
3. Known hypersensitivity or contraindication to natural or recombinant IFN-beta-1a or its excipients, or to dexamethasone or its excipients
4. Currently receiving IFN-beta-1a therapy
5. Home assisted ventilation (via tracheotomy or non-invasive) except for Continuous Positive Airway Pressure (CPAP) / Bilevel Positive Airway Pressure (BIPAP) used only for sleep-disordered breathing
6. Participation in another concurrent interventional pharmacotherapy trial during the study period
7. Decision to withhold life-sustaining treatment; patient not committed to full support (except DNR after cardiac arrest only)
8. Woman known to be pregnant, lactating or with a positive pregnancy test (urine or serum test)
9. Subject is not expected to survive for 24 hours
10. Subject has liver failure (Child-Pugh grade C)
11. Any clinical condition that in the opinion of the attending clinician or Investigator would present a risk for the subject to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Talmor, MD MPH,, Principal Investigator — Deaconess Medical Center, Spokane, Washington; Adit Ginde, MD MPH,, Principal Investigator — University of Colorado School of Medicine
Locations (4):
- United States (4):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Vanderbilt University School of Medicine, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Dexamethasone: Patients receiving active comparator: will receive two separate bolus injections one containing saline and another injection containing Dexamethasone.
  Dexamethasone: Treated daily with dexamethasone as an IV bolus for 6 days while hospitalised
Period: Overall Study
Arm/Group | IV IFN Beta-1a | IV Dexamethasone
Started | 3 | 4
Completed | 2 | 3
Not Completed | 1 | 1
Not completed — Screen Failure, patient was not dosed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV IFN Beta-1a | IV Dexamethasone | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (7.00) | 55.8 (15.69) | 57.6 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 1 | 1 | 2
  White and Other (not specified) | 0 | 2 | 2
  White | 2 | 1 | 3
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants]
  0: Able to carry out all normal activity without restriction | 3 | 3 | 6
  2: Ambulatory and capable of all self-care but unable to carry out any work activities | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Status at Day 14 (First Day of Study Drug is Day 1) as Measured by WHO 9-point Ordinal Scale
Description: WHO 9-point ordinal scale:
  0 - No detectable infection
  1. - Not hospitalized, no limitations on activities
  2. - Not hospitalized, limitation on activities
  3. - Hospitalized, not requiring supplemental oxygen
  4. - Hospitalized, requiring supplemental oxygen
  5. - Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. - Hospitalized, on invasive mechanical ventilation
  7. - Hospitalized, on mechanical ventilation plus additional organ support: renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO)
  8. - Death
Time Frame: Day 14
Population: Only 4 patients had analyzable data on D14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV IFN Beta-1a | IV Dexamethasone
Number analyzed (Participants) | 2 | 2
units on a scale | 2 (0) | 2 (0)

2. Secondary Outcome: In-hospital Mortality at Day 28 and Day 90
Description: Percentage of participants per study group that die when in still hospital at Day 28 or Day 90 of the trial
Time Frame: Day 28 and Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | IV IFN Beta-1a | IV Dexamethasone
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

3. Secondary Outcome: Overall (All-cause) Mortality at Day 28 and Day 90
Description: Percentage of participants per study group that die within 28 days or 90 days from starting the study
Time Frame: Day 28 and Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | IV IFN Beta-1a | IV Dexamethasone
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the signing of consent up to Day 28. AEs occurring after D28 were to be reported only if the Investigator considers there is a causal relationship with the study drug. All AEs up to D90, which lead to death, are reported as SAEs.
Description: All adverse events up to day 28 are reported, adverse events occurring after D28 only if the investigator considers there is a causal relationship with the study drug and all deaths up to D90.
Arm/Group | IV IFN Beta-1a | IV Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/3
Other Adverse Events (participants affected / at risk) | 1/2 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV IFN Beta-1a (N=2) | IV Dexamethasone (N=3)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV IFN Beta-1a (N=2) | IV Dexamethasone (N=3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypnoatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No formal statistical hypotheses were analysed due the early termination of the study with only 5 dosed subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT04860518/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT04860518/SAP_001.pdf